CLINICAL TRIAL: NCT00688428
Title: A Phase I, Open-Label, Randomized, Single-Center, 2-Stage Group Sequential Design, 2-Way Crossover Bioequivalence Study Comparing a Fixed-Dose Combination Capsule of Esomeprazole 40mg and Low-Dose Acetylsalicylic Acid (ASA) 325mg With a Free Combination of Esomeprazole Capsule 40mg and Low-Dose ASA
Brief Title: Study Comparing a Fixed-Dose Capsule of Esomeprazole 40mg and LDA 325mg With Free Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD, Medical Science Director NEXIUM and GI Established Brands, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: D961FC00002
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Ulcers; Upper GI Symptoms
Keywords: esomeprazole; upper gi symptoms; low dose Aspirin treatment
MeSH Terms: conditions — Ulcer | interventions — Esomeprazole; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): combination capsule of Esomeprazole 40mg + ASA 325mg
  Interventions: Drug: Esomeprazole 40mg/ASA 325mg
- 2 (Experimental): Esomeprazole 40 mg capsule and ASA 325 mg tablet
  Interventions: Drug: Esomeprazole; Drug: ASA

INTERVENTIONS:
Drug: Esomeprazole 40mg/ASA 325mg — combination capsule, administered as a single oral dose
  Other Names: Nexium/Bayer Aspirin
  Arms: 1
Drug: Esomeprazole — 40mg capsule, administered as a single dose
  Other Names: Nexium
  Arms: 2
Drug: ASA — 325mg tablet, administered as a single oral dose
  Other Names: Bayer aspirin
  Arms: 2

SUMMARY:
The purpose of this study is to test if fixed dose esomeprazole and ASA capsule is pharmaceutically equal to a free combination of esomeprazole capsule and ASA tablet

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 19-29kg/m2, inclusive
* Weight of 50-95kg, inclusive
* Clinically normal physical findings and laboratory values including hepatitis B, hepatitis C, and HIV, as judged by the Investigator

Exclusion Criteria:

* Significant clinical illness within the 2 weeks preceding the first dose of investigational products, as judged by the Investigator
* History of mental, cardiac, renal, hepatitis, neurological, or significant gastrointestinal disease, as judged by the Investigator
* Condition which could modify the absorption of the investigational products, as judged by the Investigator

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Samples for measurement of esomeprazole, ASA, and SA concentrations | Day 1 of each period

SECONDARY OUTCOMES:
Fasting blood samples for determination of clinical chemistry and hematology parameters | screening and follow up visit
urine samples for urinalysis parameters | screening, Period 1, and follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Jörgen Naesdal, M.D., Study Director — AstraZeneca; Christopher Billings ., D.O, Principal Investigator — Biokinetics Clinical Applications